CLINICAL TRIAL: NCT06511427
Title: Validation of Clinical and Ultrasonographic Scores for Prediction of Difficult Laryngoscopy and Mask Ventilation: Prospective and Evaluative Study
Brief Title: Difficult Airways Scores Validation Difficult Laryngoscopy and Mask Ventilation: Prospective and Evaluative Study
Status: Not yet recruiting | Type: Observational
Sponsor: Mongi Slim Hospital (Other)
Responsible Party: Principal Investigator, Mhamed Sami Mebazaa, Professor, Mongi Slim Hospital
Other Study IDs: difficult airway scores
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Airway Complication of Anesthesia; Ultrasound; Laryngoscopy; Difficult Airways

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- difficult laryngoscopy: patients with a cormack lehane classification after induction of anesthesia 3 or 4.
  Interventions: Diagnostic Test: upper airway sonography
- Easy laryngoscopy: patients with a cormack lehane classification after induction of anesthesia 1 or 2.
  Interventions: Diagnostic Test: upper airway sonography

INTERVENTIONS:
Diagnostic Test: upper airway sonography — clinical evaluation of upper airway, ultrasonographic assessement
  Groups: difficult laryngoscopy
Diagnostic Test: upper airway sonography — clinical evaluation of upper airway, ultrasonographic assessement
  Groups: Easy laryngoscopy

SUMMARY:
Clinical screening tests were included to define a difficult laryngoscopy such as history of difficult or impossible intubation, NC, MMS, retrognathia, protrusion of the upper incisors, TMD, mouth opening, dentition, macroglossia, presence of a beard, UBLT, spine mobility and palm print test for diabetes.

Ultrasound airway assessment was performed: Clinical screening tests were included to define a difficult laryngoscopy such as history of difficult or impossible intubation, NC, MMS, retrognathia, protrusion of the upper incisors, TMD, mouth opening, dentition, macroglossia, presence of a beard, UBLT, spine mobility and palm print test for diabetes.

Ultrasound airway assessment was performed Three parameters were measured to calculate the scores: Tongue thickness (TT) in coronal plane, Distance from the skin to hyoid bone (SHB), Distance from the skin to the thyrohyoid membrane (STM). Two scores were developed from a study conducted in 2019. The first score, to predict a difficult laryngoscopy, uses two parameters: the modified MALLAMPATI class (MMS) and the STM. A score strictly greater than 2 is predictive of a difficult laryngoscopy. The second score, to predict difficult ventilation, uses four parameters: BMI, NC, TT in coronal plane, and SHB. A score strictly greater than 20 is predictive of difficult ventilation. A well-experienced anesthesiologist performed a direct laryngoscopy and graded it as Cormack-Lehane's grading.

Difficulty in intubation and/or mask ventilation was managed according to the 2017 SFAR guidelines.

DETAILED DESCRIPTION:
The airway assessment was conducted in two phases: evaluation of clinical parameters and ultrasound parameters. Basics demographics such as age, gender, height, weight, BMI and comorbidities were noted along with the ASA classification and urgent or elective nature of the surgery. Clinical screening tests were included to define a difficult laryngoscopy such as history of difficult or impossible intubation, NC, MMS, retrognathia, protrusion of the upper incisors, TMD, mouth opening, dentition, macroglossia, presence of a beard, UBLT, spine mobility and palm print test for diabetes.

Ultrasound airway assessment was performed using a sonosite portable sonography machine with a high-frequency linear probe (10MHz) as well as a convex probe (3.5-5 MHz), with the patient lying supine and keeping the head in a neutral position. Three parameters were measured to calculate the scores: Tongue thickness (TT) in coronal plane, Distance from the skin to hyoid bone (SHB), Distance from the skin to the thyrohyoid membrane (STM). TT was measured with a low-frequency convex probe which was places submandibularly in a perpendicular plane, the cross-sectional plane was the one passing through the two lingual arteries, we considered the widest diameter. SHB was measured by placing the linear high-frequency ultrasound probe transversely over the hyoid bone. Similarly, distance from skin to the thyrohyoid membrane (STM) was measured midway between hyoid and thyroid cartilage at the level of the epiglottis.

The hyoid bone was identified as a curved echogenic structure with posterior acoustic shadow and epiglottis was identified as a curvilinear hypoechoic structure with a bright posterior air mucosal interface and hyperechoic pre-epiglottic space. Two scores were developed from a study conducted in 2019. The first score, to predict a difficult laryngoscopy, uses two parameters: the modified MALLAMPATI class (MMS) and the STM. A score strictly greater than 2 is predictive of a difficult laryngoscopy. The second score, to predict difficult ventilation, uses four parameters: BMI, NC, TT in coronal plane, and SHB. A score strictly greater than 20 is predictive of difficult ventilation. The patient was then shifted to the operating room; electrocardioscope, pulse oximetry, gas analyzer, capnography monitoring, non-invasive blood pressure, and neuromuscular blockade monitoring were connected. Other monitoring methods could be used depending on the patient condition and surgical risk, and their choice was left to the discretion of the anesthesiologist in charge of the patient. After pre-oxygenation with 100% oxygen, they were induced with intravenous injections of Sufentanil 0.3µg/kg, Propofol 3mg/kg and cisatracurium 0.15mg/kg or succinylcholine in case of a CRUSH induction. A well-experienced anesthesiologist performed a direct laryngoscopy and graded it as Cormack-Lehane's grading.

Difficulty in intubation and/or mask ventilation was managed according to the 2017 SFAR guidelines.

ELIGIBILITY:
Inclusion Criteria:

Patients aged over 18 years, scheduled for visceral or orthopedic surgery, elective or otherwise requiring general anesthesia with primary intubation and laryngoscopy, receiving a muscle relaxant before exposure were eligible for this study.

Exclusion Criteria:

Patients with conditions preventing the evaluation of clinical intubation criteria, such as altered consciousness, agitation, dementia, craniofacial or cervical spine trauma, upper areodigestive tract tumors, upper airway abnormalities or malformations, history of cervical burns or radiation therapy, thyroid goiter, tracheal stenosis, pregnancy, up to 6 weeks post-partum and situations involving extremely urgent with an immediate life- threatening prognosis as well as those undergoing intubation techniques not relying on primary laryngoscopy (e.g. optical fiberscope for mouth opening under 2.5 cm and fixed cervical spine ) were not included in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients scheduled for surgery under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-08-15 (Estimated); Primary Completion 2024-11-15 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
difficult laryngoscopy | 3 min after induction of general anesthesia
  cormack-lehane grade (from 1 to 4: 1 and 2 correspond to easy laryngoscopy and 3 or 4 to difficult laryngoscopy

SECONDARY OUTCOMES:
Difficult intubation | 3 minutes after induction of general anesthesia
  intubation requiring more than two laryngoscopies and/or the use of an alternative technique after optimizing head position (amended Jackson), with or without external laryngeal manipulation (BURP: backwards, upwards, and rightwards pressure)
Difficult mask ventilation | 3 minutes after induction of general anesthesia
  1. Inability to achieve sufficient chest expansion or a tidal volume greater than dead space (3 ml/kg), an identifiable capnographic trace, or maintain SpO2 > 92% or the Necessity to use rapid oxygen multiple times or call for another operator or the Insufflation pressure greater than 25 cmH2O;

IPD SHARING:
Plan to Share IPD: No